CLINICAL TRIAL: NCT04387448
Title: A Phase 2a Multiple Ascending, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GFB-887, a TRPC5 Channel Inhibitor, in Patients With Diabetic Nephropathy, Focal Segmental Glomerulosclerosis, and Treatment-Resistant Minimal Change Disease
Brief Title: A Study of TRPC5 Channel Inhibitor in Patients With Diabetic Nephropathy, Focal Segmental Glomerulosclerosis, and Treatment-Resistant Minimal Change Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Goldfinch Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GFB-887-201
Record Dates: First submitted 2020-05-11; First posted 2020-05-13 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Kidney Diseases; Diabetic Nephropathies; Glomerulosclerosis, Focal Segmental; Nephrosis, Lipoid; Urologic Diseases; Diabetes Complications; Diabetes Mellitus; Endocrine System Diseases; Glomerulonephritis; Nephritis; Nephrosis
MeSH Terms: conditions — Kidney Diseases; Diabetic Nephropathies; Glomerulosclerosis, Focal Segmental; Nephrosis, Lipoid; Urologic Diseases; Diabetes Complications; Diabetes Mellitus; Endocrine System Diseases; Glomerulonephritis; Nephritis; Nephrosis

STUDY DESIGN:
Intervention Model Description: Multiple-ascending, placebo-controlled
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GFB-887 multiple ascending dose (MAD) active (Experimental): GFB-887 active once-daily dosing
  Interventions: Drug: GFB-887
- GFB-887 MAD placebo (Placebo Comparator): GFB-887 placebo once-daily dosing
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GFB-887 — Investigational Medicinal Product (IMP)
  Arms: GFB-887 multiple ascending dose (MAD) active
Drug: Placebo — Matching
  Arms: GFB-887 MAD placebo

SUMMARY:
This is a phase 2a study evaluating the safety and tolerability of multiple ascending doses of GFB-887 in patients with diabetic nephropathy (DN), focal segmental glomerulosclerosis (FSGS), and treatment-resistant minimal change disease (TR-MCD).

DETAILED DESCRIPTION:
Approximately 125 patients will be enrolled in this study across the United States. Patients with DN and FSGS/TR-MCD will be randomized in 3 ascending dose cohorts to receive either GFB-887 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* All patients:

  1. Male or female 18-75 years of age, of any race, at the time of signing informed consent.
  2. Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73 m2 at Screening.
  3. Currently receiving an angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB).
* For DN patients:

  1. Diagnosis of type 2 diabetes with glycated hemoglobin (HbA1c) level ≤11% at Screening.
  2. UACR ≥ 150 mg/g.
* For FSGS/TR-MCD patients:

  1. Diagnosis of FSGS based on either biopsy or genetic testing or TR-MCD based on biopsy.
  2. UPCR ≥ 1.0 g/g.

Exclusion Criteria:

* All patients:

  1. Evidence of another (non-DN, non-FSGS/TR-MCD, respectively) kidney disease.
  2. History of malignancy, unless in remission for at least 5 years other than adequately treated basal cell or squamous cell skin cancer, cervical carcinoma in situ, or prostate cancer not expected to require treatment over the course of the study.
  3. History of any organ or bone marrow transplant, including kidney grafts.
  4. History of alcoholism or drug/chemical abuse within 12 months prior to Screening.
* For DN patients:

  1. Renal disease that requires immunosuppressive therapy (currently, or in the past).
  2. Body mass index (BMI) >45 kg/m2.
* For FSGS/TR-MCD patients:

  1. Currently on calcineurin inhibitors or history of resistance to calcineurin inhibitors.
  2. Body mass index (BMI) >40 kg/m2.
  3. Known history of severe or chronic hepatobiliary disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Percentage change in Urine Protein-to-Creatinine Ratio (UPCR) | 12 weeks
Percentage change in Urine Albumin-to-Creatinine Ratio (UACR) | 12 weeks

SECONDARY OUTCOMES:
Proportion of FSGS/TR-MCD patients achieving a modified partial remission | 12 weeks
Proportion of FSGS/TR-MCD patients achieving a complete remission | 12 weeks
Percentage change in 24-hour urine protein excretion | 12 weeks
Percentage change in 24-hour urine albumin excretion | 12 weeks
Proportion of patients (DN or FSGS/TR-MCD) with a UACR/UPCR decrease of at least 30% of baseline | 12 weeks
Proportion of patients (DN or FSGS/TR-MCD) with a UACR/UPCR decrease of at least 40% of baseline | 12 weeks
Proportion of patients (DN or FSGS/TR-MCD) with a UACR/UPCR decrease of at least 50% of baseline | 12 weeks
Incidence and severity of adverse events | 12 weeks
Incidence of clinically significant changes in 12-lead electrocardiogram (ECG) parameters, vital signs measurements, and physical examinations | Approximately 12 weeks
Incidence of clinically significant changes in laboratory parameters | 12 weeks
Plasma pharmacokinetics (PK) parameters: maximum observed plasma concentration (Cmax) | 12 weeks
Plasma PK parameters: time of the observed plasma concentration (Tmax) | 12 weeks
Plasma PK parameters: area under the plasma concentration-time curve (AUC) | 12 weeks

CONTACTS AND LOCATIONS:
Locations (74):
- United States (74):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Aventiv Research - Phoenix, Mesa, Arizona
  - Arizona Kidney Disease & Hypertension Centers (AKDHC), Scottsdale, Arizona
  - Academic Medical Research Institute (AMRI), Glendale, California
  - Amicis Research Center, Granada Hills, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Amicis Research Center, Northridge, California
  - Valley Renal Medical Group, Northridge, California
  - Respire Research - Palm Springs, Palm Springs, California
  - North American Research Institute, San Dimas, California
  - Dr. Malvin Yan Inc., South Gate, California
  - Valiance Clinical Research - Tarzana, Tarzana, California
  - Amicis Research Center, Vacaville, California
  - DaVita Mojave Sage Dialysis, Victorville, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Colorado Kidney Care (Denver Nephrology), Denver, Colorado
  - Western Nephrology - Westminster, Wheat Ridge, Colorado
  - DaVita Hartford North, Hartford, Connecticut
  - Nephrology Associationes, P.A., Newark, Delaware
  - Prohealth Research Center - Doral, Doral, Florida
  - Clinical Site Partners Leesburg, LLC, Leesburg, Florida
  - Premier Clinical Research Institute, Miami, Florida
  - Kidney & Hypertension Specialists of Miami, Miami, Florida
  - Avanza Medical Research Center, Pensacola, Florida
  - Coastal Nephrology Associates Research Center, LLC, Port Charlotte, Florida
  - Florida Premier Research Institute - Clay Street, Winter Park, Florida
  - Masters of Clinical Research, Inc., Augusta, Georgia
  - Inova Clinical Trials and Research Center, Tyrone, Georgia
  - Boise Kidney and Hypertension Institute, Meridian, Idaho
  - Research by Design, LLC, Chicago, Illinois
  - Adventist Health Partners, Hinsdale, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - University of Iowa College of Public Health, Iowa City, Iowa
  - My Kidney Center, LLC, Manhattan, Kansas
  - Louisiana Kidney Update, LLC, Lafayette, Louisiana
  - Louisiana State University Health Sciences Center - School of Medicine - New Orleans, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Renal and Transplant Associates of New England, PC, Springfield, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University School of Medicine, Detroit, Michigan
  - St. Clair Nephrology, Roseville, Michigan
  - DaVita Clinical Research, Edina, Minnesota
  - University of Minnesota - Center for Pediatric Obesity Medicine, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Nephrology & Hypertension Associates Ltd, Tupelo, Mississippi
  - Clinical Research Consultants, Kansas City, Missouri
  - DaVita Pelican Point Dialysis, Las Vegas, Nevada
  - Sierra Nevada Nephrology Consultants, Reno, Nevada
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Eastern Nephrology Associates PLLC, New Bern, North Carolina
  - Akron Nephrology Associates, Inc., Akron, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Northeast Clinical Research Center, Bethlehem, Pennsylvania
  - Rhode Island Hospital, East Providence, Rhode Island
  - South Carolina Nephrology and Hypertension, Orangeburg, South Carolina
  - Southeast Renal Research Institute, Chattanooga, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center - Amarillo, Amarillo, Texas
  - Arlington Nephrology, PC, Arlington, Texas
  - Conroe Willis Medical Research, Conroe, Texas
  - Renal Disease Research Institute, Dallas, Texas
  - El Paso Kidney Specialists, PA, El Paso, Texas
  - Xpress Trials LLC, Houston, Texas
  - Prolato Clinical Research Center, Houston, Texas
  - North Texas Kidney Disease Association, Lewisville, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - San Antonio Kidney Disease Center Physicians Group, PLLC, San Antonio, Texas
  - Clear Lake Specialties, Webster, Texas
  - Utah Kidney Research Institute, Salt Lake City, Utah
  - Tidewater Kidney Specialists - Riverview, Norfolk, Virginia
  - Providence Medical Research Center, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No